CLINICAL TRIAL: NCT00768066
Title: A Phase I/II, Randomized, Double-Blinded, Placebo-Controlled Study of the Safety and Efficacy of Transendocardial Injection of Autologous Human Cells (Bone Marrow or Mesenchymal) in Patients With Chronic Ischemic Left Ventricular Dysfunction and Heart Failure Secondary to Myocardial Infarction.
Brief Title: The Transendocardial Autologous Cells (hMSC or hBMC) in Ischemic Heart Failure Trial (TAC-HFT)
Acronym: TAC-HFT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Joshua M Hare, Director, Interdisciplinary Stem Cell Institute, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20070443
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Stem Cell Transplantation; Ventricular Dysfunction, Left
Keywords: Chronic Ischemic Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive an injection of 100 million or 200 million autologous human mesenchymal stem cells (hMSCs).
  Interventions: Biological: Autologous human mesenchymal cells (hMSCs)
- 2 (Experimental): Participants will receive an injection of 100 million or 200 million autologous human bone marrow cells (hBMCs).
  Interventions: Biological: Autologous human bone marrow cells (hBMCs)
- 3 (Placebo Comparator): Participants will receive a placebo injection of phosphate-buffered saline (PBS) and 1% human serum albumin (HAS).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Autologous human mesenchymal cells (hMSCs) — Participants will receive 40 million cells/mL delivered in either a dose of 0.25 mL per injection for a total of 1 x 108 (100 million) hMSCs x 10 injections or a dose of 0.5 mL per injection for a total of 2 x 108 (200 million) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
  Arms: 1
Biological: Autologous human bone marrow cells (hBMCs) — Participants will receive 40 million cells/mL delivered in either a dose of 0.25 mL per injection for a total of 1 x 108 (100 million) hBMCs x 10 injections or a dose of 0.5 mL per injection for a total of 2 x 108 (200 million) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
  Arms: 2
Biological: Placebo — Participants will receive 0.5 mL injections of phosphate-buffered saline (PBS) and 1% human serum albumin (HAS) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
  Arms: 3

SUMMARY:
The technique of transplanting progenitor cells into a region of damaged myocardium, termed cellular cardiomyoplasty, is a potentially new therapeutic modality designed to replace or repair necrotic, scarred, or dysfunctional myocardium. Ideally, graft cells should be readily available, easy to culture to ensure adequate quantities for transplantation, and able to survive in host myocardium; often a hostile environment of limited blood supply and immunorejection. Whether effective cellular regenerative strategies require that administered cells differentiate into adult cardiomyocytes and couple electromechanically with the surrounding myocardium is increasingly controversial, and recent evidence suggests that this may not be required for effective cardiac repair. Most importantly, transplantation of graft cells should improve cardiac function and prevent adverse ventricular remodeling. To date, a number of candidate cells have been transplanted in experimental models, including fetal and neonatal cardiomyocytes, embryonic stem cell-derived myocytes, tissue engineered contractile grafts, skeletal myoblasts, several cell types derived from adult bone marrow, and cardiac precursors residing within the heart itself. There has been substantial clinical development in the use of whole bone marrow and skeletal myoblast preparations in studies enrolling both post-infarction patients, and patients with chronic ischemic left ventricular dysfunction and heart failure. The effects of bone-marrow derived mesenchymal stem cells (MSCs) have also been studies clinically.

Currently, bone marrow or bone marrow-derived cells represent highly promising modality for cardiac repair. The totality of evidence from trials investigating autologous whole bone marrow infusions into patients following myocardial infarction supports the safety of this approach. In terms of efficacy, increases in ejection fraction are reported in the majority of the trials.

Chronic ischemic left ventricular dysfunction resulting from heart disease is a common and problematic condition; definitive therapy in the form of heart transplantation is available to only a tiny minority of eligible patients. Cellular cardiomyoplasty for chronic heart failure has been studied less than for acute MI, but represents a potentially important alternative for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ischemic left ventricular dysfunction secondary to MI.
* Be a candidate for cardiac catheterization.
* Been treated with appropriate maximal medical therapy for heart failure or post-infarction left ventricular dysfunction.
* Ejection fraction less than or equal to 50%.
* Able to perform a metabolic stress test.

Exclusion Criteria:

* Baseline glomerular filtration rate < 45 ml/min/1.73m2.
* Presence of a mechanical aortic valve or heart constrictive device.
* Documented presence of aortic stenosis (aortic stenosis graded as ≥+2 equivalent to an orifice area of 1.5cm2 or less).
* Documented presence of moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as ≥+2).
* Evidence of a life-threatening arrhythmia (nonsustained ventricular tachycardia ≥ 20 consecutive beats or complete heart block) or QTc interval > 550 ms on screening ECG. In addition; patients with sustained or a short run of ventricular tachycardia on ECG or 48 hour Ambulatory ECG during the screening period will be removed from the protocol.
* Documented unstable angina.
* AICD firing in the past 60 days prior to the procedure.
* Contra-indication to performance of a magnetic resonance imaging scan.
* Be eligible for or require coronary artery revascularization.
* Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/ul or platelet values < 100,000/ul without another explanation.
* Have liver dysfunction, as evidenced by enzymes (ALT and AST) greater than three times the ULN.
* Have a coagulopathy condition = (INR > 1.3) not due to a reversible cause.
* Known, serious radiographic contrast allergy.
* Known allergies to penicillin or streptomycin.
* Organ transplant recipient.
* Clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Non-cardiac condition that limits lifespan to < 1 year.
* On chronic therapy with immunosuppressant medication.
* Serum positive for HIV, hepatitis BsAg, or non-viremic hepatitis C.
* Female patient who is pregnant, nursing, or of child-bearing potential and not using effective birth control.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — University of Miami; Richard P Schwarz, PhD, Study Director — CV Ventures
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Result] Heldman AW, DiFede DL, Fishman JE, Zambrano JP, Trachtenberg BH, Karantalis V, Mushtaq M, Williams AR, Suncion VY, McNiece IK, Ghersin E, Soto V, Lopera G, Miki R, Willens H, Hendel R, Mitrani R, Pattany P, Feigenbaum G, Oskouei B, Byrnes J, Lowery MH, Sierra J, Pujol MV, Delgado C, Gonzalez PJ, Rodriguez JE, Bagno LL, Rouy D, Altman P, Foo CW, da Silva J, Anderson E, Schwarz R, Mendizabal A, Hare JM. Transendocardial mesenchymal stem cells and mononuclear bone marrow cells for ischemic cardiomyopathy: the TAC-HFT randomized trial. JAMA. 2014 Jan 1;311(1):62-73. doi: 10.1001/jama.2013.282909. PMID 24247587
- [Derived] Tompkins BA, Rieger AC, Florea V, Banerjee MN, Natsumeda M, Nigh ED, Landin AM, Rodriguez GM, Hatzistergos KE, Schulman IH, Hare JM. Comparison of Mesenchymal Stem Cell Efficacy in Ischemic Versus Nonischemic Dilated Cardiomyopathy. J Am Heart Assoc. 2018 Jul 12;7(14):e008460. doi: 10.1161/JAHA.117.008460. PMID 30005555
- [Derived] Trachtenberg B, Velazquez DL, Williams AR, McNiece I, Fishman J, Nguyen K, Rouy D, Altman P, Schwarz R, Mendizabal A, Oskouei B, Byrnes J, Soto V, Tracy M, Zambrano JP, Heldman AW, Hare JM. Rationale and design of the Transendocardial Injection of Autologous Human Cells (bone marrow or mesenchymal) in Chronic Ischemic Left Ventricular Dysfunction and Heart Failure Secondary to Myocardial Infarction (TAC-HFT) trial: A randomized, double-blind, placebo-controlled study of safety and efficacy. Am Heart J. 2011 Mar;161(3):487-93. doi: 10.1016/j.ahj.2010.11.024. PMID 21392602

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs): Autologous human mesenchymal cells (hMSCs): Participants will receive 40 million cells/mL delivered in a dose of 0.5 mL per injection for a total of 2 x 108 (200 million) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
- 200 Million Autologous Human Bone Marrow Cells (hBMCs): Autologous human bone marrow cells (hBMCs): Participants will receive 40 million cells/mL delivered in a dose of 0.5 mL per injection for a total of 2 x 108 (200 million) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
- Participants Will Receive a Placebo Injection of Phosphate-buf: Placebo: Participants will receive 0.5 mL injections of phosphate-buffered saline (PBS) and 1% human serum albumin (HAS) x 10 injections. The injections will be administered transendocardially during cardiac catheterization using the Biocardia Helical Infusion Catheter.
Period: Overall Study
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Started | 22 | 22 | 21
Completed | 19 | 19 | 21
Not Completed | 3 | 3 | 0
Not completed — Did not receive study product injection. | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Population: This is the number of patients who were randomized and received the study product injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf | Total
Number analyzed (Participants) | 19 | 19 | 21 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.6) | 61.1 (8.4) | 60.6 (10.4) | 59.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 18 | 17 | 20 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 9 | 26
  Not Hispanic or Latino | 11 | 9 | 12 | 32
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 16 | 18 | 20 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 21 | 59
Qualifying ejection fraction, % [Mean (Standard Deviation); unit: percent] | 35.8 (8.5) | 36.3 (11.1) | 33.0 (9.6) | 34.9 (9.7)
History of Coronary Interventions [Number; unit: participants]
  Yes | 19 | 18 | 20 | 57
  No | 0 | 1 | 1 | 2
History of Atrial/Ventricular Arrhythmia [Number; unit: participants]
  Yes | 5 | 4 | 6 | 15
  No | 14 | 15 | 15 | 44
History of Hyptertension [Number; unit: participants]
  Yes | 12 | 12 | 16 | 40
  No | 7 | 7 | 5 | 19
History of Diabetes [Number; unit: participants]
  Yes | 3 | 4 | 7 | 14
  No | 16 | 15 | 14 | 45
History of Congestive Heart Failure [Number; unit: participants]
  Yes | 11 | 16 | 16 | 43
  No | 8 | 3 | 5 | 16
History of Smoking [Number; unit: participants]
  Yes | 14 | 10 | 16 | 40
  No | 5 | 9 | 5 | 19
New York Heart Association Class [Number; unit: participants] — New York Heart Association Funcational classificaiton classifies the extent of heart failure in a patient. The 4 categories are based on how much patients are limited by physical activity, breathing, shortness of breath and/or angina pain. A class of 1 is a better New York Heart Association Class and a class of 4 is a worse New York Heart Association Class.
  participants
    I | 5 | 5 | 4 | 14
    II | 12 | 10 | 10 | 32
    III | 2 | 4 | 4 | 10
    Unknown | 0 | 0 | 3 | 3
Distance Walked in 6-Minutes [Mean (Standard Deviation); unit: meters] | 415.3 (67.9) | 399.6 (95.0) | 388.1 (58.4) | 400.6 (74.4)
Peak VO2 [Mean (Standard Deviation); unit: mL/kg/min] | 18.8 (3.8) | 17.3 (4.4) | 14.6 (5.6) | 16.7 (5.0)
Predicted FEV1 [Mean (Standard Deviation); unit: percent] | 86.2 (15.7) | 83.2 (23.2) | 79.1 (20.1) | 82.7 (19.8)
Device [Number; unit: participants] — Type of cardiac device participant had at baseline.
  participants
    Automatic implanted cardioverter-defribillator | 10 | 10 | 8 | 28
    Biventricular Pacing | 1 | 1 | 3 | 5
    None | 8 | 8 | 10 | 26
Imaging Modality [Number; unit: participants] — Type of cardiac imaging modality specified for the participant at baseline.
  participants
    MRI | 13 | 13 | 15 | 41
    CT | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence of TE-SAE Define as Composite of Death, Non-fatal MI, Stroke, Hospitalization for Worsening Heart Failure, Cardiac Perforation, Pericardial Tamponade, Ventricular Arrhythmias >15 Sec. or With Hemodynamic Compromise or Atrial Fibrillation
Time Frame: one month post-catheterization
Measure: Number; unit: participants
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
participants
  Yes | 0 | 0 | 0
  No | 19 | 19 | 21

2. Secondary Outcome: Serial Troponin Values (Every 12 Hours for the First 48 Hours Post-catheterization).
Time Frame: Measured every 12 hours for the first 48 hours post-catheterization
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
ng/mL
  Baseline | 0.06 [0.02 to 0.10] | 0.06 [0.02 to 0.11] | 0.11 [0.00 to 0.25]
  12-hours post-catheterization | 0.82 [0.47 to 1.17] | 1.03 [0.06 to 1.99] | 0.98 [0.49 to 1.47]
  24-hours post-catheterization | 0.60 [0.29 to 0.91] | 0.45 [0.04 to 0.86] | 0.42 [0.18 to 0.67]
  36-hours post-catheterization | 0.39 [0.16 to 0.62] | 0.29 [0.01 to 0.57] | 0.31 [0.13 to 0.49]
  48-hours post-catheterization | 0.31 [0.08 to 0.54] | 0.25 [0.01 to 0.49] | 0.22 [0.06 to 0.38]

3. Secondary Outcome: Serial Creatine Kinase Values (Every 12 Hours for the First 48 Hours Post-catheterization).
Time Frame: Measured every 12 hours for the first 48 hours post-catheterization
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
ng/mL
  Baseline | 1.61 [1.21 to 2.02] | 1.36 [0.80 to 1.91] | 1.64 [1.17 to 2.11]
  12-hours post-catheterization | 3.75 [2.70 to 4.80] | 2.98 [2.17 to 3.79] | 4.41 [2.31 to 6.51]
  24-hours post-catheterization | 2.19 [1.64 to 2.74] | 1.73 [1.23 to 2.24] | 2.85 [1.40 to 4.29]
  36-hours post-catheterization | 1.38 [1.11 to 1.66] | 1.28 [0.98 to 1.59] | 1.63 [1.03 to 2.23]
  48-hours post-catheterization | 1.05 [0.84 to 1.27] | 1.03 [0.79 to 1.26] | 1.36 [0.81 to 1.91]

4. Secondary Outcome: Incidence of the Major Adverse Cardiac Events (MACE) Endpoint, Defined as the Composite Incidence of (1) Death, (2) Hospitalization for Heart Failure, or (3) Non-fatal Recurrent MI.
Time Frame: 12 months post-catheterization
Measure: Number; unit: participants
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
participants
  Yes | 1 | 0 | 2
  No | 18 | 19 | 19

5. Secondary Outcome: Ectopic Tissue Formation.
Time Frame: 12 months post-catheterization
Measure: Number; unit: participants
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
participants
  Yes | 0 | 0 | 0
  No | 19 | 19 | 21

6. Secondary Outcome: Number of Deaths
Time Frame: 12-months post-catheterization
Measure: Number; unit: participants
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 19 | 19 | 21
participants
  Yes | 1 | 0 | 1
  No | 18 | 19 | 20

7. Secondary Outcome: Change From Baseline in Distance Walked in Six-minutes (Six-minute Walk Test).
Description: Data provided are with respect to the change from baseline at 12-months post-catheterization.
Time Frame: 12 months post-catheterization
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 16 | 17 | 19
meters | 32.6 [-4.6 to 69.7] | 16.9 [-14.2 to 48.0] | 6.3 [-31.4 to 44.0]

8. Secondary Outcome: Change From Baseline in the Minnesota Living With Heart Failure (MLHF) Questionnaire Total Score.
Description: Data provided are with respect to the change from baseline at 12-months post-catheterization. The Minnesota living with heart failure questionnaire uses a 6-point, zero to five, Likert scale. The total score is the sum of the 21 responses. The total score is considered the best measure of how heart failure and treatments impact a patients quality of life. The max score is 105, minimum score is 0. A lower score is considered a better quality of life.
Time Frame: 12 months post-catheterization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 16 | 17 | 15
units on a scale | -6.3 [-15.0 to 2.4] | -8.2 [-17.4 to 0.97] | 0.4 [-9.5 to 10.3]

9. Secondary Outcome: Percent Change From Baseline in Scar Mass as a Fraction of Left Ventricle Mass by Cardiac MRI or CT.
Description: Data provided are with respect to the change from baseline at 12-months post-catheterization.
Time Frame: 12 Months post-catheterization
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Number analyzed (Participants) | 14 | 15 | 16
percent change | -18.9 [-30.4 to -7.4] | -7.0 [-15.7 to 1.7] | -5.2 [-16.8 to 6.5]

ADVERSE EVENTS:
Time Frame: 30-days after transendocardial stem cell injection
Description: Adverse events are described by MedDRA preferred term.
Arm/Group | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) | Participants Will Receive a Placebo Injection of Phosphate-buf
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/19 | 3/21
Other Adverse Events (participants affected / at risk) | 6/19 | 7/19 | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) (N=19) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) (N=19) | Participants Will Receive a Placebo Injection of Phosphate-buf (N=21)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Device electrical finding (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fibrosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 Million Autologous Human Mesenchymal Stem Cells (hMSCs) (N=19) | 200 Million Autologous Human Bone Marrow Cells (hBMCs) (N=19) | Participants Will Receive a Placebo Injection of Phosphate-buf (N=21)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Investigations (Investigations) | 0 (0) | 0 (0) | 1 (1) — * Arteriogram * Electrocardiogram abnormal
Injury, Poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) — * fall * laceration * skin laceration
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) — * Dehydration * Gout
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — * Musculoskeletal pain * Myositis
Nervous system disorders (Nervous system disorders) | 1 (1) | 4 (5) | 2 (2) — * Amnesia * Dizziness * Dizziness postural * Syncope
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) — * Antiphospholipid syndrome * Splenomegaly
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) — * Dyspnoea * Pleural effusion
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) — * Pruritus * Rash
Surgical and Medical procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — - Stent placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No